CLINICAL TRIAL: NCT03394183
Title: Comparing the Efficacy of Cardiac Rehabilitation for Patients With Peripheral Artery Disease to Patients With Coronary Artery Disease
Brief Title: Efficacy of Cardiac Rehab for Patients With Peripheral Artery Disease Versus Patients With Coronary Artery Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient study personnel
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Cindy Nguyen, Principal Investigator, University Health Network, Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PVC
Record Dates: First submitted 2017-12-15; First posted 2018-01-09 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease; Coronary Artery Disease; Vascular Diseases
Keywords: cardiac rehabilitation; cardiorespiratory fitness; functional capacity; acute exercise response; quality of life
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease; Vascular Diseases | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: All participants will be enrolled in the cardiac rehabilitation program which involves weekly 1.5 hour visits at the Toronto Rehabilitation Institute Rumsey Centre for 6 months. Each visit will consist of an exercise and a risk factor education lecture. Prior to the start of the program, participants will attend two assessment sessions with cardiac rehabilitation staff members to review medical history as well as complete a cardiopulmonary exercise test. During the cardiac rehabilitation program, participants will walk at 60-80% of their VO2peak heart rate based on the results of their exercise test, as per standard care procedures. Adjustments will be made to the patient's exercise prescription under the discretion of the cardiac rehabilitation supervisor, as per standard care procedures. Patients will also be asked to exercise an additional four times during the week on their own time for a total of five times per week, as per standard care procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Artery Disease Participants (Experimental): Patients diagnosed with peripheral artery disease will undergo a 6 month cardiac rehabilitation program that is standard of care at the Toronto Rehabilitation Institute Rumsey Centre.
  Interventions: Other: Cardiac Rehabilitation
- Coronary Artery Disease Participants (Active Comparator): Patients diagnosed with coronary artery disease will undergo a 6 month cardiac rehabilitation program that is standard of care at the Toronto Rehabilitation Institute Rumsey Centre. The responses to cardiac rehabilitation for participants with coronary artery disease will be compared to participants with peripheral artery disease.
  Interventions: Other: Cardiac Rehabilitation

INTERVENTIONS:
Other: Cardiac Rehabilitation — Cardiac rehabilitation is a 6 month program in which patients enrolled attend weekly classes which consist of individualized exercise and risk factor education lectures. This intervention is consistent with standard care procedures for the Cardiovascular Prevention and Rehabilitation Program at the Toronto Rehabilitation Institute Rumsey Centre.

SUMMARY:
Exercise is commonly recommended as a treatment for patients who present with peripheral artery disease (PAD). Although a great deal of research has supported the efficacy of exercise rehabilitation for PAD, it is infrequently implemented into clinical practices.To date, no comparison of cardiac rehabilitation efficacy and acute exercise responses has been made between patients with PAD and patients with coronary artery disease (CAD). Considering some of the parallels between the two conditions, as they are both atherosclerotic conditions, and the strong recommendations for exercise in both populations, it is worthwhile to compare the efficacy of cardiac rehabilitation responses. It is also unclear if the magnitude of response for PAD patients is dependent on biological sex and clinical presentation as this may influence the development of exercise prescriptions. This study will be a prospective two-arm cohort study with both groups (CAD and PAD) undergoing the same intervention (standard 6 month out-patient cardiac rehabilitation program offered at the Toronto Rehabilitation Institute Rumsey Centre). The primary variable of interest will be peak oxygen consumption (VO2peak) with a secondary variable of interest being functional capacity, as measured by the 6-minute walk test. Tertiary variables of interest will include walking impairment, as measured by the Walking Impairment Questionnaire, and quality of life, as measured by the Short Form-36 health survey (SF-36).The second objective of this study is to determine if the magnitude of responses to cardiac rehabilitation for patients with PAD are dependent on biological sex or type of PAD (asymptomatic, post-surgical intervention, or intermittent claudication).Exploratory objectives include comparing acute exercise responses (prescribed exercise training load, actual training load, exercising heart rate and rating of perceived exertion) between PAD and CAD patients.

DETAILED DESCRIPTION:
This study is a prospective two-arm cohort study with both groups (CAD and PAD) undergoing the same intervention (standard 6 month out-patient cardiac rehabilitation program offered at the Toronto Rehabilitation Institute Rumsey Centre). The standard 6-month out-patient cardiac rehabilitation program consists of weekly 1.5 hour visits to the TRI Rumsey Centre. After determining baseline VO2peak from the exercise stress test, an individualized walking exercise prescription will be developed by a cardiac rehabilitation supervisor which corresponds to approximately 60 to 80% of the participant's VO2peak. Participants will be invited to walk around the track and attend education sessions at the same time every week for six months. Patients will be encouraged to gradually increase their exercise time walking speed. Patients will be encouraged to exercise five times a week with four sessions occurring outside of the cardiac rehabilitation program. Both PAD and CAD participants will undergo the same standard cardiac rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with lower extremity PAD or CAD
* diagnosed with concomitant PAD and CAD

Exclusion Criteria:

* vascular aneurysms, chronic heart failure, cancer, stroke, respiratory disease, or chronic kidney disease
* foot ulcers or skin breakdowns which may impede ability to exercise
* cannot follow instructions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | 6 months
  Relative VO2peak in ml/kg/min

SECONDARY OUTCOMES:
Magnitude of Response | 6 months
  To determine if the magnitude of response is dependent on biological sex or type of PAD (asymptomatic, post-surgical intervention, intermittent claudication)

OTHER OUTCOMES:
Acute Exercise Responses | 6 months
  Comparing exercising heart rate, rating of perceived exertion, and exercise prescriptions between PAD and CAD participants

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oh, Study Chair — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute Rumsey Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03394183/Prot_SAP_000.pdf